CLINICAL TRIAL: NCT05371678
Title: Comparison of Therapeutic Motor Control Interventions and Conventional Treatment in Children with Functional Constipation
Brief Title: Comparison of Two Interventions in Children with Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, nuriye ozengin, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-BI
Record Dates: First submitted 2022-04-26; First posted 2022-05-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-07

CONDITIONS: Constipation - Functional; Pediatric
Keywords: constipation; biofeedback; rehabilitation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: comparison of therapeutic motor control interventions which include education, dietary advice, core stabilization exercises, pelvic floor muscle training with surface Electromyographic, and breathing exercises and conventional treatment which include education, dietary advice and laxative therapy
Who Masked: Participant
Masking Description: Children will be divided into two intervention groups by randomization method. Randomization method will be made with a computer program (Random Allocation Software version 2.0) stratified according to age and gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic motor control interventions (Active Comparator): Treatment duration will be 8 weeks. Therapeutic motor control intervention therapy sessions will be 2 days a week. Therapeutic motor control intervention will include education about defecation and physiology, dietary advices, core stabilization exercises, pelvic floor muscle training with surface Electromyographic-Biofeedback and breathing exercises. In the first session education and dietary advices will be given to patient. Dietary advices will be given by dietitian. Two surface electromyographic electrodes will be applied on external anal sphincter muscle position.
  Interventions: Other: Therapeutic motor control interventions
- Conventional treatment (Active Comparator): Treatment duration will be 8 weeks. Conventional treatment will include education about defecation and physiology, dietary advices and laxative therapy. In the first session education and dietary advices will be given to patient. Dietary advices will be given by dietitian. Laxative therapy will be given by pediatric surgery.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Therapeutic motor control interventions — Treatment duration will be 8 weeks, two sessions a week. Each session will take approximately 60 minutes. This intervention includes education, dietary advices, core stabilization exercises and pelvic floor muscle training with surface Electromyographic-Biofeedback. In the education will be taught to the child and their parents in the first session. Dietary advices will be given by specialist dietitian. Core stabilization exercises will be performed 2 days a week with a physiotherapist and the session will be approximately 50 minutes. Diaphragmatic breathing will be taught to children in breathing exercises. The pelvic floor muscles exercises will be do by surface Electromyographic-Biofeedback. The Electromyographic-Biofeedback teaches the child how to relax the external anal sphincters with visual and auditory feedback techniques.The child will learn to relax the pelvic floor muscles during defecation by monitoring the recorded electromyographic activity.
  Arms: Therapeutic motor control interventions
Other: Conventional treatment — Treatment duration will be 8 weeks. This intervention includes education, dietary advices and laxative therapy. In the education will be taught to the child and their parents in the first session. Dietary advices will be given by specialist dietitian. Laxative therapy will be adjusted at different doses according to the child's age and weight. Laxative therapy will be administered to children by a specialist doctor.
  Arms: Conventional treatment

SUMMARY:
The purpose of this study; to compare the effects of therapeutic motor control interventions and conventional treatment in children with functional constipation on symptoms, spinal posture and mobility and trunk muscles endurance.

DETAILED DESCRIPTION:
Constipation is a very common problem in children. The pathophysiology of pediatric constipation is multifactorial and not fully understood. Constipation is a problem characterized by infrequent, difficult, often painful defecation and involuntary leakage of stool. It has been reported in the literature that the prevalence of constipation in children is 30%. It has been determined that approximately 96% of children with constipation have functional constipation.

It has been shown in the literature that children with functional constipation had a protrusion in the abdomen compared to healthy children, and their ability to actively relax their trunks decreased. Thus, it has been suggested that children with functional constipation may have reduced trunk muscle and/or endurance or muscle control. As a result of this study, they recommend that the treatment of these children should focus on awareness and education about trunk muscles, defecation and correction of sitting position.

According to the Cochrane systematic review published in 2016, physiotherapy and rehabilitation methods in bladder and bowel dysfunction are generally divided into two as education and specific methods. Specific methods are therapeutic motor control methods, manual therapy techniques (abdominal classical massage) and electrotherapy.

The use of therapeutic motor control methods in the treatment of constipation in children is quite new, and there is a need for innovative studies in this field in the literature.

The conventional treatment in children with functional constipation is education and laxatives.

In the light of this information, in this study considered that therapeutic motor control methods (core stabilization exercises, Electromyographic-Biofeedback therapy and breathing exercises) may have an effect on the symptoms of children with constipation. The primary aim of this study is to compare the effectiveness of therapeutic motor control methods and conventional treatment on constipation symptoms in children with functional constipation.

Children will be divided into 2 groups with the randomization program. Educational training, breathing exercises, dietary recommendations, core stabilization exercises and Electromyographic-Biofeedback therapy will be applied to the first group. The 2nd group is the control group and this group will receive routine treatment. Group 2 will receive laxative therapy by a specialist doctor along with educational training, dietary recommendations.

The duration of treatment will be 8 weeks. All children will be evaluated before and after 8 weeks of treatment. The first group will be treated by a physiotherapist in 2 sessions a week for 8 weeks. Each session will take approximately 60 minutes. Group 2 will receive routine treatment for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the research
* Fulfill the diagnostic criteria for functional constipation (Rome IV)

Exclusion Criteria:

* Having neurological diseases
* Having chronic diseases
* Having previous orthopedic surgery or trauma
* Presence of organic pathology underlying constipation.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Vancouver Non-Neurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome Questionnaire- symptom assessment | Eight weeks
  Vancouver Non-Neurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome Questionnaire was developed in 2009. The questionnaire consists of 14-item. Each question is 5-Likert type, and the last question is not added to the scoring. The total score ranges from 0 to 52 and increasing score means an increase in symptom severity.
7-day bowel diary (symptom assessment) | Eight weeks
  The bowel histories of the children (frequency of defecation, fecal incontinence, feeling urgency defecations...) will be evaluated with a 1-week bowel diary.

SECONDARY OUTCOMES:
Spinal Posture | Eight weeks
  Spinal posture evaluations of children will be perform with the Spinal Mouse, which is a computer-assisted and non-invasive electromechanical device. Spinal posture evaluations will be perform in standing upright position. After taking the evaluation position, the Spinal Mouse device will be moved by sliding down through all spinal processes starting from the C7 spinal process to the S3 spinal process. Relevant parameters in standing upright position [thoracic curvature angle (from T1 to T12), lumbar curvature angle (from T12 to S1), sacrum-hip angle (difference between the sacral angle and the vertical), inclination angle (angle formed by the vertical and a line joining C7 to sacrum)] were recorded by the Spinal Mouse device via bluetooth and will be analyzed.
Spinal Mobility | Eight weeks
  Spinal mobility evaluations of children will be perform with the Spinal Mouse, which is a computer-assisted and non-invasive electromechanical device. Spinal posture and mobility evaluations will be perform in 3 different positions: standing upright, maximum flexion and maximum extension. After taking the evaluation position, the Spinal Mouse device will be moved by sliding down through all spinal processes starting from the C7 spinal process to the S3 spinal process. Relevant parameters in standing upright position [thoracic curvature angle (from T1 to T12), lumbar curvature angle (from T12 to S1), sacrum-hip angle (difference between the sacral angle and the vertical), inclination angle (angle formed by the vertical and a line joining C7 to sacrum)] were recorded by the Spinal Mouse device via bluetooth and will be analyzed.
Trunk flexor muscle endurance test | Eight weeks
  In the trunk flexor endurance test, the child is in a long sitting position on the treatment bed. At this time, the trunk is supported by a wedge in 60° flexion and knees and hips flexed 90°, arms crossed in front of the chest. The feet are fixed to the bed with a belt. The wedge supporting the trunk is retracted by 10 cm and the child tries to maintain his position as much as possible. The test is terminated when the child's trunk touches the wedge or the test time exceeds 300 seconds.
Trunk extensor muscle endurance test | Eight weeks
  In the trunk extensor endurance test, the child lies in the prone position with his hips at the edge of the treatment bed. Pelvis, hips and knees are fixed to the treatment bed with belts. The child tries to keep it in a horizontal body position as much as possible by crossing his arms in front of his body. This test is terminated when the child cannot maintain the horizontal position or the test time exceeds 300 seconds.
Trunk right lateral bridge test | Eight weeks
  In the right bridge trunk endurance test, the test begins when the child's knees are extended and the upper foot is placed in front of the lower foot in the right side lying position. The child's upper arm is holding the other shoulder. The child carries his/her body weight with his/her lower elbow and feet, and he/she should keep his/her torso in a straight line as much as possible throughout the test. The test is terminated when this side lying position is disturbed or the hip touches the treatment bed or the test time exceeds 300 seconds.
Trunk left lateral bridge test | Eight weeks
  In the left bridge trunk endurance test, the test begins when the child's knees are extended and the child's upper foot is placed in front of the lower foot in the left side lying position. The child's upper arm is holding the other shoulder. The child carries his/her body weight with his/her lower elbow and feet, and he/she should keep his/her torso in a straight line as much as possible throughout the test. The test is terminated when this side lying position is disturbed or the hip touches the treatment bed or the test time exceeds 300 seconds.
Physical activity level (pedometer) | Eight weeks
  Physical activity level will be assessed by pedometer. Step counts of children will be recorded with the pedometer for a total of 4 days, 2 days on weekdays and 2 days on weekends. The pedometer will be fixed on the hips of the children.
Physical activity level (questionnaire) | Eight weeks
  Physical activity level will be assessed by questionnaire.The physical activity questionnaire for children (PAQ-C) will assess physical activity the ages of 8-14 years.The total score of the PAQ-C consists of the first 9 items. A score of 1 means low level of physical activity, while a score of 5 means high physical activity. PAQ for Adolescents (PAQ-A) is a questionnaire designed to evaluate the physical activity of students aged 14-20 attending secondary education during the last 7 days of the school term.A score of '1' corresponds to low-intensity physical activity and a score of '5' corresponds to high-intensity physical activity, but the last question is not included in the scoring. The total score is obtained by calculating the average score of all questions.
Evaluation of subjective perception of improvement | Eight weeks
  The Global Perceived Impact scale will be used to evaluate children after treatment (week 8). Children will be asked to rate the extent to which their complaints have improved on a 4-item Likert-type scale. Description of scores; '1' would be 'worsened', '2' would be 'unchanged', '3' would be 'better', '4' would be 'completely healed'
Evaluation of compliance with lifestyle changes | Eight weeks
  After the treatment (8th week), the degree of compliance of the children with the recommendations for lifestyle changes will be evaluated with the Visual Analog Scale. Children will be asked to mark the point that best describes them on a vertical line 10 cm long. The distance of the marked point to the '0' point will be measured with a ruler and recorded in cm. On this scale, the '0' point will be defined as 'Never (0%) I Have Not Complied' and the '10' point will be defined as 'I Have Fully (100%) Compliance'.
Evaluation of compliance with breathing exercises | Eight weeks
  After the treatment, the degree of compliance of the children in Group 1 towards breathing exercises will be evaluated with the Visual Analog Scale. Children will be asked to mark the point that best describes them on a vertical line 10 cm long. The distance of the marked point to the '0' point will be measured with a ruler and recorded in cm. On this scale, the '0' point will be defined as 'Never (0%) I Have Not Complied' and the '10' point will be defined as 'I Have Fully (100%) Compliance'.

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Ozengin, Ph.D., Principal Investigator — Bolu Abant İzzet Baysal University; Büşra İnal, M.Sc., Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No